CLINICAL TRIAL: NCT03912675
Title: Role of Autologous Dermal Micrografts in Regenerative Surgery
Brief Title: Dermal Micrografts in Regenerative Surgery
Acronym: Rigenera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2142CE
Record Dates: First submitted 2019-04-04; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Regenerative Medicine
Keywords: Cell transplants; Autografting

STUDY DESIGN:
Intervention Model Description: The study includes 20 patients with 24 post-surgical defect in any site of the body with a size range 4-400 cm2. The acute post-surgical soft tissue loss is considered the experimental unit of the study irrespective of the number of wounds per patient. Each unit is randomized to be treated either with Integra® dermal substitute enriched with the autologous dermal micro-grafts obtained with RigeneraTM protocol (group A - RigeneraTM protocol - 12 units) or with Integra® dermal substitute only (group B - Control - 12 units). The expected endpoint is a spontaneous re-epithelialization higher than 25% of the total wound area in group A at 4 weeks. The secondary endpoint is the comparison of the re-epithelialization rate at 4 weeks after the first surgical stage between the group A and the controls. The re-epithelialization rate in the wounds is assessed through digital photography with the software "Image J".
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RigeneraTM protocol (Experimental): Teatment with Integra® dermal substitute enriched with the autologous dermal micro-grafts obtained with RigeneraTM protocol.
  Interventions: Procedure: Integra® dermal substitute and RigeneraTM protocol
- Control (Experimental): Treatment with Integra® dermal substitute only.
  Interventions: Procedure: Integra® dermal substitute and RigeneraTM protocol

INTERVENTIONS:
Procedure: Integra® dermal substitute and RigeneraTM protocol — Integra® dermal substitute enriched with the autologous dermal micro-grafts obtained with RigeneraTM protocol

SUMMARY:
Objective assessment of the effectiveness of a micro-fragmented dermal extract obtained with Rigenera™ technology (patented by Human Brain Wave) in promoting the wound healing process in an in-vivo homogeneous experimental human acute surgical wound model.

DETAILED DESCRIPTION:
The aim of the study is the objective assessment of the effectiveness of a micro-fragmented dermal extract obtained with Rigenera™ technology (patented by Human Brain Wave) in promoting the wound healing process in an in-vivo homogeneous experimental human acute surgical wound model. The study includes 20 patients with 24 acute post-surgical soft tissue loss and a planned sequential two-stage repair with dermal substitute and autologous split-thickness skin graft. Each acute post-surgical soft tissue loss is randomized to be treated either with Integra® dermal substitute enriched with the autologous dermal micro-grafts obtained with Rigenera™ technology (group A - Rigenera™ protocol) or with Integra® dermal substitute only (group B - Control). The re-epithelialization rate in the wounds is assessed in both groups at 4 weeks through digital photography with the software "Image J". The dermal cell suspension enrichment with the Rigenera™ technology is considered effective if the re-epithelialized area is higher than the 25% of the total wound surface as this threshold is considered far beyond the expected spontaneous re-epithelialization rate.

ELIGIBILITY:
Inclusion Criteria:

* Post-surgical defect in any site of the body with a size range 4-400 cm2.

Exclusion Criteria:

* Wound infection, chemotherapy in the last 6 months, use of corticosteroids or immunosuppressive treatment, metabolic, endocrine, autoimmune and collagen diseases.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Spontaneous re-epithelialization. | 4 weeks
  Percentage of patients with spontaneous re-epithelialization of the total wound surface higher than 25% as assessed by Image J Software

CONTACTS AND LOCATIONS:
Overall Officials: Angela Faga, Professor, Principal Investigator — Università degli Studi di Pavia
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy

REFERENCES:
- [Derived] Tresoldi MM, Graziano A, Malovini A, Faga A, Nicoletti G. The Role of Autologous Dermal Micrografts in Regenerative Surgery: A Clinical Experimental Study. Stem Cells Int. 2019 Sep 8;2019:9843407. doi: 10.1155/2019/9843407. eCollection 2019. PMID 31582991